CLINICAL TRIAL: NCT03196375
Title: A Randomized, Double-Blind, Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of FLX-787-ODT for Treatment of Muscle Cramps in Adult Subjects With Motor Neuron Disease
Brief Title: A Study to Assess FLX-787 in Subjects With Motor Neuron Disease Experiencing Muscle Cramps.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor
Sponsor: Flex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLX-787-203
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Motor Neuron Disease
Keywords: Motor Neuron Disease; Neurodegenerative Diseases; Nervous System Diseases; Neuromuscular Diseases; Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Progressive Muscular Atrophy; Muscle cramps; Muscle cramping; ALS; MND; PMA; PLS; FLX-787
MeSH Terms: conditions — Motor Neuron Disease; Neurodegenerative Diseases; Nervous System Diseases; Neuromuscular Diseases; Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Muscle Cramp; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: FLX-787-ODT (orally disintegrating tablet)
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo ODT

INTERVENTIONS:
Drug: FLX-787-ODT (orally disintegrating tablet) — FLX-787-ODT taken three times daily for 28 days
  Arms: Experimental
Drug: Placebo ODT — Placebo ODT taken three times daily for 28 days
  Arms: Placebo Comparator

SUMMARY:
The COMMEND Study will assess the safety and effectiveness of FLX-787 in men and women with Motor Neuron Disease [including Amyotrophic Lateral Sclerosis (ALS), Primary Lateral Sclerosis (PLS) or Progressive Muscular Atrophy (PMA)] experiencing muscle cramps. Participants will be asked to take two study products during the course of the study. One of these study products will be a placebo.

Approximately 120 participants in approximately 30 study centers across the United States are expected to take part. Participants will be in the study for approximately 3 months and visit the study clinic 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Motor Neuron Disease (MND) [including Amyotrophic Lateral Sclerosis (ALS), Primary Lateral Sclerosis (PLS) or Progressive Muscular Atrophy (PMA)]
* Expected survival > 6 months
* Weekly muscle cramping (defined as: a sustained muscle contraction that's most often painful and lasts seconds to minutes)

Exclusion Criteria:

* Presence of major gastrointestinal disorders, such as inflammatory bowel disease, diverticulitis, active peptic ulcer disease, or significant gastroesophageal reflux disease (i.e., not well-controlled on antacids or proton pump inhibitors), or oral or esophageal lesions/ulcers
* Presence of laryngospasm or significant swallowing problems
* Presence of percutaneous endoscopic gastrostomy, esophagogastroduodenoscopy, or G-tube
* Unable or unwilling to discontinue medications for cramps and/or opiates
* Inability to tolerate a spicy sensation in the mouth or stomach
* Actively using illicit drugs or history of chronic substance abuse within the past year prior to screening, including abuse of alcohol
* Intention to change the current level of tobacco use or use of nicotine-containing products (i.e., new smokers or those actively trying to quit may not enrolled)
* Participated in a clinical study (except natural history studies without administration of an investigational product) within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Cramp frequency | 28 days
  Cramp frequency measured over the 28-day treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Oskarsson, MD, Principal Investigator — Mayo Clinic Jacksonville Florida
Locations (35):
- United States (35):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - California Pacific Medical Center, Sacramento, California
  - University of California - Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - GW Medical Faculty Associates Inc., Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida Health, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Neuroscience Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Providence Brain and Spine Institute, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Neuromuscular Center, Austin, Texas
  - Baylor Scott and White Health, Round Rock, Texas
  - UT Health San Antonio, San Antonio, Texas
  - The University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Saint Luke's Rehabilitation Institute, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided